CLINICAL TRIAL: NCT04488991
Title: Naboth Kisti ve HPV pozitifliği arasındaki ilişkinin araştırılması
Brief Title: Nabothian Cyst Protects or Facilitates Against Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Cihan Comba, gynecological oncology specialist, Haseki Training and Research Hospital
Other Study IDs: 2020-74
Record Dates: First submitted 2020-07-16; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: HPV Infection; Nabothian Cyst; Cervical Cancer
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cervical swap samples will be used as Biospecimen to get know whether there is HPV infection in cervix, and which tipe of HPV infection occurs in patients' cervix
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- the woman who has just HPV infection: the woman who is between 30-65 years old, who is participate this research, and has just HPV infection in cervix.
  Interventions: Other: Cervical Cancer Rate
- the woman who has just nabothian cyst: the woman who is between 30-65 years old, who is participate this research, and has just nabothian cyst in cervix.
  Interventions: Other: Cervical Cancer Rate
- the woman who has both nabothian cyst and HPV infection: the woman who is between 30-65 years old, who is participate this research, and has both nabothian cyst in cervix.
  Interventions: Other: Cervical Cancer Rate

INTERVENTIONS:
Other: Cervical Cancer Rate — In the end of the Research, we will compare cervical cancer rates between groups

SUMMARY:
Aim of the study to asses the realition between HPV infection, Nabothian Cyst and Cervical Intraepithelial lesions or Cervical Cancer

DETAILED DESCRIPTION:
Nabothian cysts are one of the common gynecological pathologies. They rarely have clinical significance. Transvaginal ultrasonography and magnetic resonance imaging are the most useful imaging methods for cervical cystic lesions.HPV infection is the most important factor which can cause cervical malignancy and premalignant lesions. In women between 30-65 years of age HPV-DNA testing, is used as a screening test in Turkey. In this research, the aim is to examine whether there is a connection between Naboth cysts and HPV infection in the cervix. During the examination, the swab sample required for HPV PCR testing will be taken. The number and size of Naboth cysts with vaginal USG will be noted. If the patient had colposcopy / LEEP (Loop Electrosurgical Excision Procedure), the result will be investigated and noted.

ELIGIBILITY:
Inclusion Criteria:

To have Naboth cyst and/or HPV positivity Must be willing and able to provide informed consent Comply with the study protocol Between 25-65 age range

Exclusion Criteria:

To Refuse participate in our research The age under 25 and over 65 Ovarian, endometrial and vulvar malignancies Without both Naboth's cyst and HPV positivity To have LEEP/Cervical Conization before History of Cervical Dysplasia

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: the woman; who is between 25-65 years of age, who goes to Haseki Education and Research Hospital Gynecology and Oncology Outpatient Clinic, who has nabothian cyst and/ or HPV infection
Sampling Method: Non-Probability Sample
Enrollment: 1005 (Estimated)
Dates: Start 2020-07-23 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Nabothian cyst affects the HPV infection in cervix | through study completion, an average of 1 year
  in the research, results will be compared for to figure out the relation; nabothian cyst how affects HPV infection , how causes cervical dysplasia in cervix.

SECONDARY OUTCOMES:
Does the other factors(like cigarette, birth number, vaginitis) affect HPV infection and Cervical Cancer | through study completion, an average of 1 year
  In the research Other factors(like cigarette, birth number, vaginitis) will be also noted. These datas will be used to understand correlation; the other factors increase or decreate the rate of HPV infection and cervical dysplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Cihan Comba, MD, Study Chair — Sultangazi Haseki Training and Research Hospital
Locations (1):
- Cihan Comba, Istanbul, Sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malagon T, Volesky KD, Bouten S, Laprise C, El-Zein M, Franco EL. Cumulative risk of cervical intraepithelial neoplasia for women with normal cytology but positive for human papillomavirus: Systematic review and meta-analysis. Int J Cancer. 2020 Nov 15;147(10):2695-2707. doi: 10.1002/ijc.33035. Epub 2020 May 26. PMID 32363604
- [Background] Isoda T, BaBa S, Maruoka Y, Kitamura Y, Nishie A, Sasaki M, Honda H. Nabothian cyst a predominant cause of false-positive iodine uptake in uterus: comparison of SPECT/CT and pelvic MRI. Clin Nucl Med. 2014 Aug;39(8):680-4. doi: 10.1097/RLU.0000000000000504. PMID 24978344
- [Result] Barrigon A, Ziadi S, Jacot-Guillarmod M, Da Silva S, Dumont M, Raineri I, Bongiovanni M. Nabothian cyst content: A potential pitfall for the diagnosis of invasive cancer on Pap test cytology. Diagn Cytopathol. 2019 Feb;47(2):127-129. doi: 10.1002/dc.24098. Epub 2018 Oct 24. PMID 30353714
- [Result] D'Alessandro P, Giudicepietro A, Della Corte L, Arduino B, Saccone G, Iacobelli A, Insabato L, Zullo F. A case of gastric-type mucinous endocervical adenocarcinoma in presence of nabothian cysts. Eur J Obstet Gynecol Reprod Biol. 2019 May;236:254-255. doi: 10.1016/j.ejogrb.2019.02.024. Epub 2019 Mar 2. No abstract available. PMID 30878235